CLINICAL TRIAL: NCT05660304
Title: Modulating Language Networks in Patients With Post-stroke Aphasia Using Cortico-cortical Paired Associative Stimulation
Brief Title: Studying Language With Brain Stimulation in Aphasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Julio C Hernandez Pavon, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00217734
Record Dates: First submitted 2022-11-09; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Stroke; Aphasia
Keywords: Transcranial Magnetic Stimulation; Stroke Aphasia; Language; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Stroke; Aphasia; Language

STUDY DESIGN:
Intervention Model Description: A parallel randomized study will be performed. Three patients will be randomly assigned to receive ccPAS followed by speech-language therapy or sham ccPAS followed by speech-language therapy. Whether the participant receives ccPAS or sham ccPAS alongside speech-language therapy will be determined, at random, using a randomized number generator and enrollment order.
Who Masked: Participant
Masking Description: Because of the nature of the study, study personnel administering brain stimulation cannot be masked regarding whether the participant receives ccPAS or sham ccPAS. To minimize bias, neither the participant nor the speech-language pathologist will have knowledge of which group the participant is assigned to. However, the researcher administering ccPAS or sham ccPAS will know which intervention is applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ccPAS group (Experimental): Patients under this group will receive ccPAS followed by speech-language therapy.
  Interventions: Device: Cortico-cortical paired associative stimulation
- Sham ccPAS group (Sham Comparator): Patients under this group will receive sham ccPAS followed by speech-language therapy.
  Interventions: Device: Sham cortico-cortical paired associative stimulation

INTERVENTIONS:
Device: Cortico-cortical paired associative stimulation — Two brain areas will be stimulated with transcranial magnetic stimulation pulses. The pulses will be delivered with a time difference, on other words, one pulse after another.
  Arms: ccPAS group
Device: Sham cortico-cortical paired associative stimulation — Two brain areas will be stimulated with sham transcranial magnetic stimulation. The sham pulses will be delivered with a time difference, on other words, one pulse after another.
  Arms: Sham ccPAS group

SUMMARY:
The overall goal of this study is to evaluate whether stimulation of two brain areas alongside behavioral speech-language therapy increases connectivity to improve language functions in stroke-aphasia patients.

DETAILED DESCRIPTION:
The brain is made up of networks that communicate with each other to help us think and communicate. After a stroke, networks between different areas of the brain can lose connection. In the case of aphasia, networks in the language areas of the brain are often disrupted. There is currently no "fix" to restore these specific language connections. However, transcranial magnetic stimulation (TMS) might help the areas reconnect through alternative pathways.

TMS is a non-invasive procedure (in other words, it takes place outside your body). A coil will be placed over your head. The coil sends magnetic pulses to your brain to stimulate, or excite, neurons. Most studies using TMS stimulate one area of the brain at a time, but this does not tell us how to improve the network connections between brain areas.

For this study, we plan to stimulate two language areas of the brain to improve these network connections. To do this, we will use a form of TMS called "cortico-cortical paired associative stimulation" (ccPAS). This type of TMS involves applying paired pulses to two different brain areas that have been "disconnected" from each other after a stroke. The pulses are delivered with a time difference, on other words, one pulse after another.

If you choose to participate, you will be randomly assigned to one of two groups. There is a 50% chance you will receive active brain stimulation with speech-language therapy and a 50% chance that you will receive inactive or sham stimulation (no brain stimulation) along with speech-language therapy. Neither you nor the clinician on the research project will choose - or know - which group you are assigned to. Only the person administering the stimulation will know.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of non-fluent aphasia due to a single, left-hemisphere stroke
2. ≧ six months post-stroke onset
3. WAB-R Fluency, Grammatical Competence, and Paraphasias Score between 2-6
4. 18+ years of age
5. Premorbidly right-handed
6. English-speaking
7. Ability to participate in fMRI / TMS protocol

Exclusion Criteria:

1. Cardiac pacemaker or pacemaker wires; neurostimulators; implanted pumps
2. Metal in the body (rods, plates, screws, shrapnel, dentures, IUD) or metallic particles in the eye
3. Surgical clips in the head or previous neurosurgery
4. Any magnetic particles in the body
5. Cochlear implants
6. Prosthetic heart valves
7. Epilepsy or any other type of seizure history
8. History of significant head trauma (i.e., extended loss of consciousness, neurological sequelae)
9. Significant other disease (heart disease, malignant tumors, mental disorders)
10. Significant claustrophobia
11. Ménière's disease
12. Medications that increase risk of seizures, for instance antipsychotic and antidepressant medications acting primarily on the central nervous system, which lower the seizure threshold such as antipsychotic drugs (chlorpromazine, clozapine) or tricyclic antidepressants
13. Non-prescribed drug use, for instance recreational marijuana
14. Unable to refrain from using any alcohol and nicotine products for at least 24 hours before the study Visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-09 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in functional connectivity with resting-state functional magnetic resonance imaging (rs-fMRI) | Before vs. after ccPAS/sham ccPAS, on Days 1, 5, and 10 of the ccPAS/sham ccPAS regimen. We also compare the responses from Day 1 vs. Day 10.
  A seed-based functional connectivity analysis will be carried out between the two stimulated brain areas. To assess the changes in effective connectivity, we will compare the seed-based connectivity values across sessions.

SECONDARY OUTCOMES:
Changes in the Western Aphasia Battery-Revised (WAB-R) Reading subtest | Visit 1 (baseline, pre-intervention), Visit 12 (immediately post-intervention), and Visit 13 (maintenance, 1-month post-intervention).
  The WAB-R Reading subtest will be administered to assess changes in overall reading ability pre- and post-intervention as well as at the 1-month follow-up.
Changes in oral reading probes | Visit 3 (baseline, pre-intervention), Visit 7 (midpoint, of intervention), Visit 12 (immediately post-intervention), and Visit 13 (maintenance, 1-month post-intervention).
  Oral reading probes will be administered to assess changes in oral reading of trained and untrained sentence stimuli before/after intervention session 1, after intervention session 5, before/after intervention session 10, and at the 1-month follow-up.
Changes on The Short-Form Philadelphia Naming Test (PNT) | Visit 3 (baseline, pre-intervention), Visit 12 (immediately post-intervention), and Visit 13 (maintenance, 1-month post-intervention).
  The Short-Form Philadelphia Naming Test (PNT) will be administered to assess changes in overall naming ability before/after intervention session 1, before/after intervention session 10, and at the 1-month follow-up.
Changes in production of connected speech using standardized expositional discourse stimuli (Broken Window and Cat in Tree picture scenes) | Visit 3 (baseline, pre-intervention), Visit 12 (immediately post-intervention), and Visit 13 (maintenance, 1-month post-intervention).
  Discourse elicitation tasks (e.g., picture descriptions) will be administered to assess changes in overall discourse ability (e.g., correct information units, rate) before/after intervention session 1, before/after intervention session 10, and at the 1-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Julio Hernandez Pavon, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No